CLINICAL TRIAL: NCT00803647
Title: A Phase II Study to Determine the Surgical Conversion Rate in Patients Receiving Neoadjuvant mFOLFOX7 + Cetuximab for Unresectable Wild-Type K-RAS Colorectal Cancer With Metastases Confined to the Liver
Brief Title: A Study With Neoadjuvant mFOLFOX7 Plus Cetuximab to Determine the Surgical Conversion Rate for Unresectable Colorectal Cancer With Metastases Confined to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-6
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2016-09-14 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: NSABP; Cetuximab; FOLFOX7; Oxaliplatin; Leucovorin; 5-FU; colorectal cancer; KRAS wild type; metastatic colorectal cancer; Erbitux; Eloxatin; Liver resection; Liver ablation; Metastasectomy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): mFOLFOX7 (5-FU, leucovorin, oxaliplatin) + cetuximab
  Interventions: Biological: cetuximab; Drug: 5-FU; Drug: oxaliplatin; Drug: leucovorin

INTERVENTIONS:
Biological: cetuximab — 500 mg/m2 IV every two weeks on days 1, 15, 29, and 43 of each 56 day cycle, for a total of 3 cycles. Cetuximab dose will be escalated by 100 mg/m2 every 2 weeks to a maximum dose of 800 mg/m2 if, at the time of retreatment, skin rash is less than or equal to grade 1, diarrhea is grade 0 (defined as less than or equal to 3 stools per day over baseline), and the patient is not experiencing any other greater than or equal to grade 2 toxicity attributed to cetuximab.
  Other Names: Erbitux
Drug: 5-FU — 3000 mg/m2 IV continuous infusion over 46 hours every two weeks on days 1, 15, 29, and 43 of each 56 day cycle, for a total of 3 cycles.
  Other Names: 5-fluorouracil
Drug: oxaliplatin — 85 mg/m2 IV every two weeks on days 1, 15, 29, and 43 of each 56 day cycle, for a total of 3 cycles.
  Other Names: Eloxatin
Drug: leucovorin — 400 mg/m2 IV every two weeks on days 1, 15, 29, and 43 of each 56 day cycle, for a total of 3 cycles.

SUMMARY:
FC-6 is a Phase II, multi-center clinical trial for patients with unresectable, wild-type K-RAS, colorectal cancer with metastases confined to the liver. Liver metastases must be determined by FC-6 criteria to be unresectable, and the colorectal cancer (CRC) tumor (primary or metastatic) must be found to be wild-type K-RAS. Patients with mutant K-RAS tumors are ineligible. K-RAS testing can be done through the local hospital or a tumor sample can be submitted to the FC-6 central lab (Esoterix Clinical Trial Services).

A primary aim of this study is to evaluate the surgical conversion rate using cytotoxic combination chemotherapy and biologic therapy with cetuximab, a monoclonal antibody targeted against the epidermal growth factor receptor. A second primary aim is to evaluate the safety and tolerability of a chemotherapy/targeted therapy regimen in this patient population. Secondary aims include determination of clinical response rate, recurrence-free survival for patients undergoing complete resection and/or ablation of liver metastases, and overall survival.

DETAILED DESCRIPTION:
All patients will receive the FC-6 study treatment regimen every 2 weeks during each 8-week cycle for a total of 3 cycles.

Baseline imaging of the chest, abdomen, and pelvis will be performed. CT scan or MRI of the abdomen will be performed after 1 cycle of neoadjuvant therapy to assess clinical response and resectability of liver metastases. If liver metastases are not deemed to be resectable at this assessment, but tumor assessment demonstrates stable disease or partial response, therapy will continue with re-assessment for clinical response and resectability after Cycle 2 and, if necessary, after Cycle 3.

After a minimum of 1 cycle of therapy, patients who meet the guidelines for resection of liver metastases will undergo liver metastasectomy (tumor resection and/or ablation) as soon as judged technically feasible by the hepatic surgeon in order to minimize chemotherapy damage to the liver and morbidity from surgery. At the investigator's discretion, the chemotherapy and cetuximab regimen may be continued for 1 additional treatment given at least 2 weeks before the planned date of surgery. This additional treatment, if given, will not be considered to be part of the 3 study therapy cycles.

The surgical goal is to perform a curative (R0) resection and/or ablation. If curative surgery was performed and if only 1 or 2 cycles of therapy were administered before surgery, postoperative therapy using the same regimen will resume 4-6 weeks following surgery to complete 3 cycles of study treatment. Following discontinuation of study therapy, all patients who undergo R0 resection (with or without ablation) will be followed every 3 months for the first 2 years on the study and then every 6 months for years 3 through 5.

Further therapy for patients who do not undergo R0 resection/ablation will be at the investigator's discretion. These patients will only be followed for vital status every 12 months for the remainder of the 5-year period following study entry.

A total sample size of 60 patients will be enrolled in the FC-6 trial.

ELIGIBILITY:
Conditions for patient eligibility

* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and must be considered a potential candidate for a major hepatic surgical procedure.
* The patient must have histologic or cytologic confirmation of a diagnosis of colorectal adenocarcinoma.
* There must be documentation by PET/CT scan, CT scan, MRI, or intraoperative palpation (at the time of resection of the primary colorectal tumor, if applicable) that the patient has evidence of hepatic metastasis. (Histologic confirmation of hepatic metastasis is not required.)
* Patients are eligible with any of the following: primary tumor and regional nodes resected with clear surgical margins and no evidence of extrahepatic disease or; unresected primary tumor with plans to resect the primary tumor prior to study entry or; unresected primary tumor with plans to resect the primary tumor and the liver metastases in a single surgical procedure performed within 2-7 weeks after the last preoperative dose of chemotherapy/cetuximab or; unresected primary with plans to resect the primary tumor and the liver metastases in staged procedures performed within 2-7 weeks after the last preoperative dose of chemotherapy/cetuximab.
* The colorectal primary tumor or metastatic tumor must be determined to be wild-type K-RAS. The K-RAS test may have been performed through the local hospital, or a tumor sample may be submitted to the FC-6 central lab for K-RAS testing. If local K-RAS test results are reported as indeterminate, submission of a tumor sample for central testing is required. Note: Needle biopsy of liver metastasis is not recommended for the express purpose of obtaining tissue for K-RAS testing because of the risk of needle track dissemination of malignant cells.
* There must be documentation that the liver metastases must have been determined by a hepatic surgeon approved (by protocol defined criteria) to participate in FC-6 to be unresectable based on at least one of the following criteria: All of the liver metastases cannot be resected (and/or ablated) with negative margins, i.e., lesion(s) located in an area that would result in the resection of all of the hepatic veins or the main portal vein or the right and left hepatic arteries or the common bile duct; Complete resection and/or ablation would require greater than 60% of the liver parenchyma to be removed. Note: At the discretion of the hepatic surgeon, portal vein embolization (PVE) may be utilized preoperatively following neoadjuvant therapy to enhance the volume of the hepatic remnant. However, the determination of unresectability will be based on the estimate, at the time of study entry, of the percentage of liver parenchyma that would need to be removed. PVE may be employed preoperatively to enhance the overall safety, but not specifically the resectability of the liver metastasis(es).
* There must be documentation that: at least 3 of the 8 hepatic segments are free of metastases or; based on imaging studies, the patient is anticipated to have at least 40% of the liver will remain intact after surgery.
* If an adjuvant therapy regimen of 5-FU given alone or in combination with leucovorin, irinotecan, capecitabine, oxaliplatin, cetuximab, or bevacizumab was administered, the adjuvant therapy must have been discontinued more than 6 months prior to study entry.
* The patient must have had the following tests and exams within 4 weeks prior to study entry: medical history and physical exam; consultation with a hepatic surgeon approved for FC-6; and PET/CT scan or both a PET scan and a CT scan of the chest, abdomen, and pelvis must be performed. (MRI scan can be substituted for the CT scan.)
* There must be evidence of adequate bone marrow function: absolute neutrophil count (ANC) greater than or equal to 1500/mm3; Hemoglobin greater than or equal to 10 g/dL; Platelets greater than or equal to 100,000/mm3
* There must be evidence of adequate hepatic function: Total bilirubin less than or equal to upper limit of normal (ULN) for the lab; aspartate aminotransferase (AST) less than or equal to 5.0 x ULN for the lab
* Serum creatinine must be less than or equal to 1.5 mg/dL.

Conditions for patient ineligibility

* Diagnosis of anal or small bowel carcinoma.
* Colorectal cancers other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.
* Unresected primary tumor in the colon or rectum with significant symptoms related to obstruction or that will require radiation therapy.
* Evidence of extrahepatic metastases or non-contiguous extension of intrahepatic metastases to non-hepatic tissues.
* Radiographic evidence of metastases to portal lymph nodes (node greater than 1 cm in diameter) unless the node(s) are proven by biopsy to be negative.
* Previous hepatic resection and/or ablation, hepatic arterial infusion therapy, or any systemic therapy for metastatic disease. (Patients who have only had an excisional biopsy are eligible.)
* Radiation therapy to the liver.
* Pre-existing chronic hepatic disease (e.g., chronic active hepatitis, cirrhosis) that, in the opinion of the investigator and hepatic surgeon, would limit the patient's ability to undergo hepatic metastasectomy.
* Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 grade 3 or 4 anorexia or nausea related to metastatic disease.
* CTCAE v3.0 greater than or equal to grade 2 vomiting related to metastatic disease.
* CTCAE v3.0 greater than or equal to grade 2 sensory/motor neuropathy.
* Any of the following cardiac conditions: Documented congestive heart failure; Myocardial infarction within 6 months prior to study entry; Unstable angina within 6 months prior to study entry; Symptomatic arrhythmia.
* Serious or non-healing wound, skin ulcers, or bone fracture.
* History of bleeding diathesis or coagulopathy. (Patients on stable anticoagulant therapy are eligible.)
* Symptomatic interstitial lung disease or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients.
* Any evidence of active infection.
* Active inflammatory bowel disease.
* Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, colorectal carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Previous serious hypersensitivity reaction to monoclonal antibodies.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Pregnancy or lactation at the time of study entry. (WOCBP must have a negative pregnancy test within 2 weeks prior to study entry. Male and female patients of reproductive potential must agree to use adequate contraceptive methods during and for 2 months after study therapy. )
* Any other serious concomitant medical condition that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to participate in the study.
* Use of any investigational product within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (23):
- United States (23):
  - Loma Linda University Medical Center, Loma Linda, California
  - St. Joseph Hospital, Orange, California
  - Kaiser Permanente-San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - CCOP - NorthShore University HealthSystem, Evanston, Illinois
  - Edward Hospital, Naperville, Illinois
  - University of Iowa, Iowa City, Iowa
  - NortonHealthcare, Inc., Louisville, Kentucky
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP, William Beaumont Hospital, Royal Oak, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP, Dayton, OH, Dayton, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - NSABP Foundation, Inc., Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.4)
Sex/Gender, Customized [Number; unit: participants] | NA — Gender data were not collected.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Had a Curative (R0) Liver Metastasectomy Following Protocol Treatment, i.e., Metastatic Disease That Can be Completely Resected and/or Ablated With no Postoperative Evidence of Residual Malignant Disease (R0 Resection).
Time Frame: 8 months
Population: All 20 patients were included in this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
percentage of participants | 75 [50.9 to 91.34]

2. Primary Outcome: Reported Adverse Events.
Description: 19 participants experienced at least one adverse event. There were a total of 95 adverse events reported. (Note: multiple occurrences of the same adverse event in one individual are counted only once.) Refer to the Adverse Events section for specifics. The Other Adverse Events section lists only those events occurring above 5% frequency.
Time Frame: 8 months
Measure: Number; unit: adverse events
Arm/Group | Treatment
Number analyzed (Participants) | 20
adverse events | 95

3. Secondary Outcome: Overall Survival (OS). Time From Study Entry Until Death From Any Cause.
Description: The percentage of patients alive at 18 months.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
percentage of participants | 83.8 [57.7 to 94.5]

4. Secondary Outcome: Objective Clinical Response Rate (cRR). Measureable Lesions That Can be Accurately Measured in at Least One Dimension With Conventional Radiologic Techniques or Spiral CT.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by PET/CT, CT scan, MRI or spiral CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective clinical Response Rate (cRR) = CR + PR during the 3 preoperative cycles, among the treated patients.
Time Frame: 8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
percentage of participants | 85 [62.1 to 96.8]

5. Secondary Outcome: Recurrence-free Survival (RFS). Time From Study Entry Until First Recurrence.
Time Frame: 2 years
Population: Patients with R0 resection
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 15
months | 13.3 [5.5 to 23.2]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
septic shock (Infections and infestations) | 1 (1)
wound infection (Infections and infestations) | 1 (1)
vascular access complication (Injury, poisoning and procedural complications) | 2 (2)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 1 (1)
arhythmia supraventricular (Cardiac disorders) | 1 (1)
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
thrombosis in device (General disorders) | 1 (1)
hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
platelet count decreased (Investigations) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1)
venous thrombosis (Vascular disorders) | 1 (1)
Cavernous sinus thrombosis (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
alanine aminotransferase increased (Investigations) | 2 (2)
aspartate aminotransferase increased (Investigations) | 2 (2)
blood alkaline phosphatase increased (Investigations) | 2 (2)
exfoliative rash (Skin and subcutaneous tissue disorders) | 6 (6)
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 7 (7)
anaemia (Blood and lymphatic system disorders) | 3 (3)
leukopenia (Blood and lymphatic system disorders) | 3 (3)
lymphopenia (Blood and lymphatic system disorders) | 2 (2)
decreased appetitie (Metabolism and nutrition disorders) | 2 (2)
hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
fatigue (General disorders) | 2 (2)
hypersensitivity (Immune system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days